CLINICAL TRIAL: NCT04465552
Title: Arrhythmic Manifestations and Management Strategies in Hospitalized COVID-19 Patients: Proposal for a Multicenter Registry
Brief Title: Arrhythmic Manifestations and Management in Hospitalized COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRF-COVID-19-0001
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infections
Keywords: COVID-19; Arrhythmic Manifestations; Management Strategies
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized COVID-19 Patients
  Interventions: Other: Patients received standard of care treatment during hospitalization

INTERVENTIONS:
Other: Patients received standard of care treatment during hospitalization — All patients admitted with covid-19 will be enrolled and followed for the duration of their hospitalization as well as during outpatient follow for up to 6 months, in those recovered, to assess clinical outcomes.

SUMMARY:
Although arrhythmias appear to be common in COVID-19 patients, arrhythmia mechanisms and characteristics, predisposing factors, incidence of sudden cardiac death and predictors, therapeutic strategies employed as well as long term outcomes are not well understood. Hence, we seek to develop a multicenter registry aimed to characterize arrhythmic manifestations, employed treatment strategies and long-term outcomes among hospitalized COVID-19 patients in the US.

DETAILED DESCRIPTION:
The novel coronavirus (SARS-CoV-2) and the resulting respiratory tract infection (Coronavirus Disease 2019 or COVID-19) is a pandemic with over 3 million cases globally and resulting in >230,000 deaths at the time of this writing. From initial reports in Wuhan, China, viral progression resulted in over 80,000 cases in January/February 2020 in China. The following global spread has involved more than 210 countries. Unfortunately, the United States has been significantly affected, with over 1 million confirmed cases and over 60,000 deaths, the highest in the world. As this global pandemic continues to rage, cardiovascular, especially arrhythmic manifestations associated with COVID-19 have become evident. A recent report from Wuhan, China, noted that 16.7% of hospitalized and 44.4% of ICU patients with COVID-19 had arrhythmias. Although arrhythmias appear to be common in COVID-19 patients, arrhythmia mechanisms and characteristics, predisposing factors, incidence of sudden cardiac death and predictors, therapeutic strategies employed as well as long term outcomes are not well understood. Hence, we seek to develop a multicenter registry aimed to characterize arrhythmic manifestations, employed treatment strategies and long-term outcomes among hospitalized COVID-19 patients in the US.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Hospital admission with COVID-19

Exclusion Criteria:

● Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Hospitalized COVID-19 patients > 18 years of age
Sampling Method: Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
To better characterize arrhythmic manifestations, employed treatment strategies and long- term outcomes in hospitalized COVID-19 patients in the US through a multicenter retrospective chart review. | January 1, 2020 - June 30, 2020
  To better characterize arrhythmic manifestations, employed treatment strategies and long- term outcomes in hospitalized COVID-19 patients in the US through a multicenter retrospective chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Gopinathannair, MD, Principal Investigator — Kansas City Heart Rhythm Research Foundation
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. "Coronavirus Cases." Worldometer, www.worldometers.info/coronavirus/. Accessed March 28, 2020.
- [Background] 2. "Covid-19 Interactive Map." Johns Hopkins Coronavirus Resource Center, 2020, coronavirus.jhu.edu/map.html. Accessed March 28, 2020.
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] 4. Centers for Disease Control and Prevention. Interim Clinical Guidance for Management of Patients with Confirmed 2019 Novel Coronavirus (2019-nCoV) Infection, https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinical-guidance-management-patients.html
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076